CLINICAL TRIAL: NCT06640491
Title: Intraosseous Vancomycin and Cefazolin vs Intravenous Administration in Primary Total Knee Arthroplasty
Brief Title: Intraosseous (IO) Cefazolin and Vancomycin in Primary Total Knee Arthroplasty (TKA)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Brian Parsley, Physician, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00038477
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraosseous Administration of Vancomycin and Cefazolin (Experimental): Intraosseous vancomycin plus cefazolin is administered via an intraosseous cannulation device (Arrow EZ-IO; Teleflex, Morrisville, NC) in the OR after sterile prep of the leg and draping has occurred prior to skin incision and after the tourniquet has been inflated. The injection will take place into the tibial tubercle, which is a known safe IO injection site. The IO injection will include 500mg of vancomycin and a 1g dose of cefazolin, previously used in prior IO studies of cefazolin.
  Interventions: Drug: IO Administration of Cefazolin; Drug: IO Administration of Vancomycin
- Standard IV Administration of Vancomycin and Cefazolin (Active Comparator): Patients will receive the Houston Methodist Hospital orthopedic surgery standard of care pre-operative antibiotic regimen for primary total knee arthroplasty patients. This includes IV antibiotics cefazolin will be started in the pre-operative period approximately 1 hour prior to incision. The cefazolin dose is generally 2g if patient is under 120kg, and 3g is the patient is above 120kg in line with guidelines. Vancomycin IV administration will be dosing will be weight-based at approximately 15mg/kg generally 1000-1750mg in 500mL NS.
  Interventions: Drug: IV Administration of Cefazolin; Drug: IV Administration of Vancomycin

INTERVENTIONS:
Drug: IO Administration of Cefazolin — Intraosseous injection of cefazolin to guard against infection.
  Arms: Intraosseous Administration of Vancomycin and Cefazolin
Drug: IO Administration of Vancomycin — Intraosseous injection of vancomycin to guard against infection.
  Arms: Intraosseous Administration of Vancomycin and Cefazolin
Drug: IV Administration of Cefazolin — Intravenous dose of cefazolin to guard against infection.
  Arms: Standard IV Administration of Vancomycin and Cefazolin
Drug: IV Administration of Vancomycin — Intravenous dose of vancomycin to guard against infection.
  Arms: Standard IV Administration of Vancomycin and Cefazolin

SUMMARY:
The goal of this clinical trial is to compare the efficacy of intravenous (IV) and intraosseous (IO) antibiotic administration techniques during primary total knee arthroplasty (TKA) in adults undergoing a TKA procedure at Houston Methodist Hospital. The main questions it aims to answer are:

Does IO administration of vancomycin and cefazolin protect against perioperative exposure risks? Is there a difference in post-operative complication rates between IV and IO administration of these drugs?

Participants will be randomized to receive either the standard of care IV administration of Vancomycin and Cefazolin, or the IO administration of Vancomycin and Cefazolin.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to undergo an elective primary total knee arthroplasty.
* Patient is able to understand the study design and intervention and gives informed consent to participate in the study.
* Patient is 18 years or older.

Exclusion Criteria:

* Contraindication to receiving vancomycin or cefazolin.
* Body mass index (BMI) > 40.
* Uncontrolled Diabetes (defined as A1c > 7.5%).
* Patient received or is scheduled to receive IV vancomycin or cefazolin within 7 days prior to their planned procedure.
* Any hardware, condition, or anatomic status that prevents the tibial tubercle from being a viable intraosseous injection site.
* Refusal to participate
* Any condition, in the opinion of the primary investigator, that deems the participant unsuitable for participation in the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Infections | 30 days postop and 90 days postop
  Participants charts will be reviewed at 30 days postop and 90 days postop to determine if there were any infections.

SECONDARY OUTCOMES:
Postoperative Wound Complications | 30 days postop and 90 days postop
  Participants charts will be reviewed at 30 days postop and 90 days postop to determine if there were any wound complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nunn MO, Corallo CE, Aubron C, Poole S, Dooley MJ, Cheng AC. Vancomycin dosing: assessment of time to therapeutic concentration and predictive accuracy of pharmacokinetic modeling software. Ann Pharmacother. 2011 Jun;45(6):757-63. doi: 10.1345/aph.1P634. Epub 2011 Jun 7. PMID 21652786
- [Background] Klasan A, Patel CK, Young SW. Intraosseous Regional Administration of Vancomycin in Primary Total Knee Arthroplasty Does Not Increase the Risk of Vancomycin-Associated Complications. J Arthroplasty. 2021 May;36(5):1633-1637. doi: 10.1016/j.arth.2020.12.034. Epub 2020 Dec 26. PMID 33468344
- [Background] Parkinson B, McEwen P, Wilkinson M, Hazratwala K, Hellman J, Kan H, McLean A, Panwar Y, Doma K, Grant A. Intraosseous Regional Prophylactic Antibiotics Decrease the Risk of Prosthetic Joint Infection in Primary TKA: A Multicenter Study. Clin Orthop Relat Res. 2021 Nov 1;479(11):2504-2512. doi: 10.1097/CORR.0000000000001919. PMID 34397615
- [Background] Park KJ, Chapleau J, Sullivan TC, Clyburn TA, Incavo SJ. 2021 Chitranjan S. Ranawat Award: Intraosseous vancomycin reduces periprosthetic joint infection in primary total knee arthroplasty at 90-day follow-up. Bone Joint J. 2021 Jun;103-B(6 Supple A):13-17. doi: 10.1302/0301-620X.103B6.BJJ-2020-2401.R1. PMID 34053300
- [Background] Chin SJ, Moore GA, Zhang M, Clarke HD, Spangehl MJ, Young SW. The AAHKS Clinical Research Award: Intraosseous Regional Prophylaxis Provides Higher Tissue Concentrations in High BMI Patients in Total Knee Arthroplasty: A Randomized Trial. J Arthroplasty. 2018 Jul;33(7S):S13-S18. doi: 10.1016/j.arth.2018.03.013. Epub 2018 Mar 15. PMID 29655497
- [Background] Young SW, Zhang M, Freeman JT, Mutu-Grigg J, Pavlou P, Moore GA. The Mark Coventry Award: Higher tissue concentrations of vancomycin with low-dose intraosseous regional versus systemic prophylaxis in TKA: a randomized trial. Clin Orthop Relat Res. 2014 Jan;472(1):57-65. doi: 10.1007/s11999-013-3038-z. PMID 23666589
- [Background] Harper KD, Lambert BS, O'Dowd J, Sullivan T, Incavo SJ. Clinical outcome evaluation of intraosseous vancomycin in total knee arthroplasty. Arthroplast Today. 2020 Mar 7;6(2):220-223. doi: 10.1016/j.artd.2020.02.001. eCollection 2020 Jun. PMID 32577466
- [Background] Young SW, Zhang M, Freeman JT, Vince KG, Coleman B. Higher cefazolin concentrations with intraosseous regional prophylaxis in TKA. Clin Orthop Relat Res. 2013 Jan;471(1):244-9. doi: 10.1007/s11999-012-2469-2. PMID 22773397
- [Background] Von Hoff DD, Kuhn JG, Burris HA 3rd, Miller LJ. Does intraosseous equal intravenous? A pharmacokinetic study. Am J Emerg Med. 2008 Jan;26(1):31-8. doi: 10.1016/j.ajem.2007.03.024. PMID 18082778
- [Background] Petitpas F, Guenezan J, Vendeuvre T, Scepi M, Oriot D, Mimoz O. Use of intra-osseous access in adults: a systematic review. Crit Care. 2016 Apr 14;20:102. doi: 10.1186/s13054-016-1277-6. PMID 27075364
- [Background] de Lalla F, Novelli A, Pellizzer G, Milocchi F, Viola R, Rigon A, Stecca C, Dal Pizzol V, Fallani S, Periti P. Regional and systemic prophylaxis with teicoplanin in monolateral and bilateral total knee replacement procedures: study of pharmacokinetics and tissue penetration. Antimicrob Agents Chemother. 1993 Dec;37(12):2693-8. doi: 10.1128/AAC.37.12.2693. PMID 8109937
- [Background] Yamada K, Matsumoto K, Tokimura F, Okazaki H, Tanaka S. Are bone and serum cefazolin concentrations adequate for antimicrobial prophylaxis? Clin Orthop Relat Res. 2011 Dec;469(12):3486-94. doi: 10.1007/s11999-011-2111-8. Epub 2011 Oct 4. PMID 21968901
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Background] Sivagnanam S, Deleu D. Red man syndrome. Crit Care. 2003 Apr;7(2):119-20. doi: 10.1186/cc1871. Epub 2002 Dec 23. PMID 12720556
- [Background] Feder OI, Yeroushalmi D, Lin CC, Galetta MS, Meftah M, Lajam CM, Slover JD, Schwarzkopf R, Bosco JA 3rd, Macaulay WB. Incomplete Administration of Intravenous Vancomycin Prophylaxis is Common and Associated With Increased Infectious Complications After Primary Total Hip and Knee Arthroplasty. J Arthroplasty. 2021 Aug;36(8):2951-2956. doi: 10.1016/j.arth.2021.03.035. Epub 2021 Mar 18. PMID 33840539
- [Background] Classen DC, Evans RS, Pestotnik SL, Horn SD, Menlove RL, Burke JP. The timing of prophylactic administration of antibiotics and the risk of surgical-wound infection. N Engl J Med. 1992 Jan 30;326(5):281-6. doi: 10.1056/NEJM199201303260501. PMID 1728731
- [Background] Peel TN, Astbury S, Cheng AC, Paterson DL, Buising KL, Spelman T, Tran-Duy A, Adie S, Boyce G, McDougall C, Molnar R, Mulford J, Rehfisch P, Solomon M, Crawford R, Harris-Brown T, Roney J, Wisniewski J, de Steiger R; ASAP Trial Group. Trial of Vancomycin and Cefazolin as Surgical Prophylaxis in Arthroplasty. N Engl J Med. 2023 Oct 19;389(16):1488-1498. doi: 10.1056/NEJMoa2301401. PMID 37851875
- [Background] Liu C, Kakis A, Nichols A, Ries MD, Vail TP, Bozic KJ. Targeted use of vancomycin as perioperative prophylaxis reduces periprosthetic joint infection in revision TKA. Clin Orthop Relat Res. 2014 Jan;472(1):227-31. doi: 10.1007/s11999-013-3029-0. PMID 23645338
- [Background] Burger JR, Hansen BJ, Leary EV, Aggarwal A, Keeney JA. Dual-Agent Antibiotic Prophylaxis Using a Single Preoperative Vancomycin Dose Effectively Reduces Prosthetic Joint Infection Rates With Minimal Renal Toxicity Risk. J Arthroplasty. 2018 Jul;33(7S):S213-S218. doi: 10.1016/j.arth.2018.03.009. Epub 2018 Mar 14. PMID 29656981
- [Background] Siddiqi A, Forte SA, Docter S, Bryant D, Sheth NP, Chen AF. Perioperative Antibiotic Prophylaxis in Total Joint Arthroplasty: A Systematic Review and Meta-Analysis. J Bone Joint Surg Am. 2019 May 1;101(9):828-842. doi: 10.2106/JBJS.18.00990. PMID 31045673
- [Background] Spangehl M. Preoperative Prophylactic Antibiotics in Total Hip and Knee Arthroplasty: What, When, and How. J Arthroplasty. 2022 Aug;37(8):1432-1434. doi: 10.1016/j.arth.2022.01.019. Epub 2022 Jan 17. PMID 35051610
- [Background] Ahmed SS, Haddad FS. Prosthetic joint infection. Bone Joint Res. 2019 Dec 3;8(11):570-572. doi: 10.1302/2046-3758.812.BJR-2019-0340. eCollection 2019 Nov. No abstract available. PMID 31832177
- [Background] Rodriguez-Merchan EC, Delgado-Martinez AD. Risk Factors for Periprosthetic Joint Infection after Primary Total Knee Arthroplasty. J Clin Med. 2022 Oct 18;11(20):6128. doi: 10.3390/jcm11206128. PMID 36294449
- [Background] Mortazavi SM, Schwartzenberger J, Austin MS, Purtill JJ, Parvizi J. Revision total knee arthroplasty infection: incidence and predictors. Clin Orthop Relat Res. 2010 Aug;468(8):2052-9. doi: 10.1007/s11999-010-1308-6. PMID 20309657
- [Background] Koh CK, Zeng I, Ravi S, Zhu M, Vince KG, Young SW. Periprosthetic Joint Infection Is the Main Cause of Failure for Modern Knee Arthroplasty: An Analysis of 11,134 Knees. Clin Orthop Relat Res. 2017 Sep;475(9):2194-2201. doi: 10.1007/s11999-017-5396-4. Epub 2017 Jun 1. PMID 28573549